CLINICAL TRIAL: NCT03933514
Title: Metagenomic and Immune-inflammatory Analysis of Individuals With Generalized Aggressive Periodontitis and Their Descendants.
Status: Completed | Type: Observational
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Renato Casarin, Professor Dr., University of Campinas, Brazil
Other Study IDs: 079/2013
Record Dates: First submitted 2019-04-29; First posted 2019-05-01 (Actual); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Generalized Aggressive Periodontitis
Keywords: Family; Microbiome; Cytokines; Aggressive Periodontitis
MeSH Terms: conditions — Aggressive Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Dental Biofilm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- GAgP parents: Parents diagnosed with Generalized Aggressive Periodontitis
- GAgP children: Children from parents diagnosed with Generalized Aggressive Periodontitis
  Interventions: Other: Plaque control
- Health parents: Parents diagnosed as periodontally healthy
- Health children: children from parents diagnosed as periodontally healthy
  Interventions: Other: Plaque control

INTERVENTIONS:
Other: Plaque control — Children were instructed about the hygiene procedures
  Groups: GAgP children; Health children

SUMMARY:
Generalized aggressive periodontitis (GAgP) is a multifactorial disease related to several aspects that influence its installation and progression. A constant microbial colonization, an altered inflammatory response, and a clear genetic factor are cited as possible factors associated with this pathology. Thus, aggressive periodontitis subjects could transmit for their descendants some genetical alterations, such as inflammatory response pattern associated with periodontal destruction and susceptibility to colonization by some pathogens, increasing the risk of develops this disease. This way, this project is aimed to evaluate the pattern of microbiological colonization and the inflammatory response pattern associated with it, comparing parents with generalized aggressive periodontitis and their children and periodontally healthy parents and their children. Thirty families will be selected and divided into two groups: Test group (n=15 families) families in which the parents (or at least one of them) present generalized aggressive periodontitis and one child (age ranging from 6-12 years old); Control group (n=15 families) families in which the parents (both of them) present periodontal healthy and one child (age ranging from 6-12 years old). The groups will be composed using a gender- and age-matched structure. The children will participate in a hygiene program and will be monitored for 3 months. All individuals (parents and children) will be clinically assessed for plaque and bleeding index, periodontal probing depth, clinical attachment level and gingival recession. During this period, samples of gingival crevicular fluid (GCF) and subgingival biofilm from periodontal pockets/sites from all subject (parents and children) will be collected. The GCF will be analyzed and the detection of interleukin (IL)-1β, IL-4, IL-6, IL-8, IL-10, IL-17, tumor necrosis factor (TNF)-α, and interferon (INF)-γ will be done using Luminex/MAGpix technology. In a subgingival biofilm, the DNA will be extracted and the microbiome and its functional characteristics will be evaluated by metagenomics and bioinformatics analysis. The data will be compared by Student's t-test, Mann-Whitney e Wilcoxon tests. The significance level for all analysis will be 5%.

ELIGIBILITY:
Inclusion Criteria:

* GAgP parents: i) less than 35 years old at the diagnosis; ii) at least 8 teeth with probing depth (PD) and clinical attachment level (CAL) > 5mm (with at least 2 sites with PD > 7mm) at diagnosis; iii) at least 20 teeth in the oral cavity; iv) good systemic health.
* Health parents: i) Good systemic health; ii) at least 20 teeth in the oral cavity; iii) absence of periodontal pockets/gingival sulcus with PD > 4mm; iv) absence of proximal bone loss.
* Children: i) to present parents respecting the inclusion criteria for periodontal health or GAgP; ii) 6 to 12 years of age at the beginning of study iii) good systemic health iv) presence of first molars and central incisors.

Exclusion Criteria

* the use of antibiotics and anti-inflammatory medication 6 months prior to the study;
* smoking habits
* pregnancy or lactation.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The population selected from Piracicaba Dental School graduation clinic
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Change of the baseline plaque index on probing at 3 months | Baseline and 3 months for each test
  Reduction in the amount of plaque accumulation around the gingival marginal after the therapy.

SECONDARY OUTCOMES:
Change of the baseline bleeding on probing at 3 months | Baseline and 3 months for each test
  Bleeding induced at the depth of the gingival sulcus or periodontal pocket after probing
Change of the baseline inflammatory markers levels in gingival crevicular fluid (pg/uL) at 3 months | Baseline and 3 months for each test
  Concentration of IL-1β, IL-4, IL-6, IL-8, IL-10, IL-17, TNF-α and INF-γ released in gingival crevicular fluid
Change in the microbial composition at 3 months | Baseline and 45 days for each test
  Concentration of bacteria in the subgingival biofilm

IPD SHARING:
Plan to Share IPD: Undecided